CLINICAL TRIAL: NCT05117606
Title: ABLY LYNG Study at Helse More Romsdal - Aalesund Sykehus HMR With the Ably LYNG Patient Care Solution Advanced Prototype by Ably Medical AS.
Brief Title: LYNG21: Ably LYNG Clinical Demonstration in Operative Environment
Acronym: LYNG21
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Ably Medical AS (Industry)
Collaborators: Alesund Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LYNG21_AALESUND
Record Dates: First submitted 2021-09-14; First posted 2021-11-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-10

CONDITIONS: Monitoring, Physiologic
Keywords: non-intrusive monitoring

STUDY DESIGN:
Intervention Model Description: Within subject comparison - of two screening methodologies (standard equipment with direct patient sensors vs LYNG contactless sensors). The number patients in the study is chosen to have a broad view on patients population found in a general hospital setting, for example a range of height, weight, gender, age.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vitalsigns (Other): Data from patients (heart rate, respiration, movement, blood pressure) is measured with traditional, standard hospital equipment in parallell with data from LYNG mat captured non-intrusively in the same session.
  Interventions: Device: LYNG by Ably Medical

INTERVENTIONS:
Device: LYNG by Ably Medical — Comparing LYNG to traditional, standard equipment for heart rate, respiration, movement, and blood pressure.

SUMMARY:
The study main objective will be to compare measurements of heart rate, respiration rate, blood pressure and movement done by LYNG by Ably Medical with the corresponding measurements made by standard equipment in a patient sample in a hospital setting. The comparison will show the degree of agreement between LYNG and the existing current standard equipment. Data from the study will support Ably Medical in optimizing the LYNG product and measurement precision.

DETAILED DESCRIPTION:
The LYNG sensor mat is placed beneath a regular bed matrass and captures data without direct patient contact. Data collected by the LYNG sensor is transmitted via cables to the bed-side connectivity box for initial local analysis and storage. Data will be extracted and formatted for post-analysis in additional software for verification and validation purposes.

Specifically, the LYNG study objectives are as follows:

1. collect sensor data from LYNG Solution to optimize the LYNG data algorithms to further improve parameter estimations of patient heart rate, respiratory rate, blood pressure and movement indicators.
2. Compare parameter estimation by LYNG against current and relevant standard of care measurement methods

The study design is a within-subjects comparison in parameter estimation with Ably LYNG as comparator to standard of care. Patients will take part in 60-minute sessions where measurements are collected in accidence to standard procedure for the standard equipment while the LYNG system collects the same data non- intrusively. The data will not be part of any clinical decision making or have any impact of the patient care. The study will take place during Q2-Q3/2021 with estimated 8-12 weeks duration including logistics, setup, data collection, study closure.

ELIGIBILITY:
Inclusion Criteria:

* For patients:

  * Admitted to hospital,
  * Able to provide voluntary, informed consent.

Exclusion Criteria:

* For patients:

  * Health condition that endangers patient by participation due to pain, rehabilitation, and/or negative impact on treatment or care, as evaluated by medical personnel,
  * Pregnancy,
  * Significantly reduced mobility that implies substantial strain for moving in and out of bed, as evaluated by medical personnel
  * Unable to provide informed, voluntary consent personally or by legal guardian, * below 18 years old,
  * Patients with implantable devices such as pacemakers, baclofen pumps, insulin pumps, etc, or
  * Any way identified as 'vulnerable'

The nurse handing recruitment will explicitly check for inclusion/exclusion criteria alignment and document this in the study Enrolment Form. The routine will be to check for formal criteria and to describe the study in such a manner that the patient understands content, and make sure the patient understands before consenting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-05-25 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Absolute Relative Error of Heart Rate (beats per minute) | 60 minutes
  absolute relative error = (reference measure/LYNG measure)/Reference
Absolute Relative Error of Respiration Rate (respirations per minute) | 60 minutes
  absolute relative error = (reference measure/LYNG measure)/Reference
Movement | 60 minutes
  Comparison of movement as part of patient instruction compared to indications of movement in movement sensors. Qualitative analysis.
absolute relative error of Blood Pressure = (reference measure/LYNG measure)/Reference | 60 minutes
  absolute relative error = (reference measure/LYNG measure)/Reference
  Sphygmomanometer, millimeters of mercury (mmHg) upper (systolic), lower (diastolic), and mean value.

CONTACTS AND LOCATIONS:
Overall Officials: Dag A Lihaug Hoff, Principal Investigator — HMR Aalesund Hospital
Locations (1):
- Helse Møre og Romsdal HF - Aalesund Sjukehus, Ålesund, Norway